CLINICAL TRIAL: NCT05577988
Title: Assessment of an Early De-Escalation to a Low-potency Single Antiplatelet Therapy Guided by Genetics Versus a Systematic High-Potency Single Antiplatelet Therapy to Neutralize Bleeding Complications in Patients With High Bleeding Risk Beyond One Month After an Acute Coronary Syndrome
Acronym: ADEN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fonds de Dotation ACTION (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: APHP211027; 20-0570 PHRC (Other: DGOS)
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: MYOCARDIAL INFARCTION
Keywords: Acute Coronary Syndrome; High Bleeding Risk; Antiplatelet Therapy
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: National, multicentre, comparative, controlled, randomized, open label trial using the PROBE study design (Prospective Randomized Open Blinded End-point)
Who Masked: Outcomes Assessor
Masking Description: Members of the Endpoint Adjudication Committee (AEC) are blinded to randomization group, treatments and characteristics.
  The Committee will assess all endpoints according to the definitions stated in the protocol. This will be a blinded evaluation. Clinical endpoint adjudication will be performed using blinded source data that are provided by CRAs to the committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Standard of Care : Systematic de-escalation to a high potency antiplatelet single therapy
- Intervention arm (Other): single-antiplatelet with a low-potency antiplatelet (aspirin or clopidogrel) guided by genetic testing.
  Interventions: Other: single-antiplatelet with a low-potency antiplatelet (aspirin or clopidogrel) guided by genetic testing.

INTERVENTIONS:
Other: single-antiplatelet with a low-potency antiplatelet (aspirin or clopidogrel) guided by genetic testing. — * Individuals without genetic loss of function to metabolize clopidogrel (*1/*1, *2/*17, *3/*17): stop DAPT and switch to a single antiplatelet therapy by clopidogrel.
  * Individuals with genetic loss of function to metabolize clopidogrel (*2/*3, 1/*3, *2/*2, *1/*2,*3/*3): stop potent P2Y12 inhibitor and treat with a single antiplatelet therapy by aspirin.
  * Individuals with fast metabolization of clopidogrel (*1/*17 or *17/*17): stop potent P2Y12 inhibitor and treat with a single antiplatelet therapy by aspirin.
  Arms: Intervention arm

SUMMARY:
Patients who suffered from acute coronary syndrome (ACS) are usually treated with a long-term dual antiplatelet therapy (DAPT) to reduce stent thrombosis and recurrent ischemic event. Nonetheless, recent important data have demonstrated the efficacy of a short term DAPT and an early single antiplatelet therapy in high bleeding and ischemic risk patients.

The bleeding risk is associated with a significant mortality. This risk is especially high in patients treated with potent P2Y12 inhibitors like ticagrelor or prasugrel after an ACS.

As a result of the abounding data regarding the safety of an early single antiplatelet therapy with high potency antiplatelet therapy (ticagrelor or prasugrel), it is likely that such strategy will soon be implemented in the guidelines.

The benefits of these high-potency P2Y12 inhibitors over clopidogrel mostly occur in patients with genetic polymorphisms of CYP2Y12 associated with a loss of function in clopidogrel metabolism.

Furthermore, the anti-ischemic benefit of potent P2Y12 inhibitors over clopidogrel occurs early, while excess bleeding events often arise during chronic treatment.

Our hypothesis is that a systematic and rapid genetic screening of CYP2C90 *2 or *17 polymorphism to guide an early single therapy with low potency antiplatelet (aspirin or clopidogrel) could lead to less bleeding events with a consistent efficacy towards cardiac events compared with high potency antiplatelet therapies (prasugrel or ticagrelor) in high bleeding risk patients treated for ACS.

DETAILED DESCRIPTION:
Multicenter, randomized, open label trial using the PROBE study design. Randomization 1 to 3 months (preferably 1, considering the HBR) after ACS into 2 parallel arms. Stratification: according to revascularization status (PCI or no PCI), genotype (loss of function, fast metabolization, none) and center.

Control arm: stop aspirin for a single antiplatelet therapy with a high-potency antiplatelet (ticagrelor or prasugrel).

Intervention arm: single-antiplatelet with a low-potency antiplatelet (aspirin or clopidogrel) guided by genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* Being 18-year-old or older
* Admission for type 1 acute myocardial infarction (STEMI or NSTEMI)
* Bedside genetic testing for clopidogrel resistance that can be performed during hospital stay for ACS (oral swab kit with result within 1 hour)
* Treated with aspirin and ticagrelor, or aspirin and prasugrel at the screening phase and at the randomization visit.
* High bleeding risk as defined below (criteria adapted from the Consensus Document From the Academic Research Consortium for High Bleeding Risk) (at least one criterion) :

  * Age ≥75 years old.
  * Baseline haemoglobin <11 g/dl (or anaemia requiring transfusion during the 4 weeks prior to randomization).
  * Chronic Kidney Disease with estimated glomerular filtration rate ≤ 30 ml/min.
  * Thrombocytopenia with platelet count < 100 x 109 / L
  * Chronic bleeding diatheses: inherited or acquired conditions known to be associated with increased bleeding risk such as platelet dysfunction, von Willebrand disease (prevalence of 1%-2% in the general population), inherited or acquired clotting factor deficiencies (including factors VII, VIII [hemophilia A], IX [hemophilia B], and XI), or acquired antibodies to clotting factors, among others.
  * Cirrhosis with portal hypertension.
  * PCI after major traumatism or surgery.
  * Any documented stroke in the last 12 months.
  * Hospital admission for bleeding or transfusion within last 6 months.
  * Nonskin cancer diagnosed or treated ≤3 years.
  * Planned daily nonsteroidal anti-inflammatory drugs (other than aspirin) or steroids for ≥30 days after PCI.
* patient affiliated to a social security system
* signed informed consent form
* Women of childbearing capacity with effective contraception for the duration of the research OR man, OR woman not of childbearing capacity

Exclusion Criteria:

* Currently participating in any interventional investigational device or drug trial
* Any prior documented intracerebral bleed
* Contra-indication, known allergy or expected interactions with clopidogrel. Baseline treatment (at screening) should not include an antiplatelet therapy for which a contra-indication, known allergy or expected interactions is known (example history of stroke and use of prasugrel, or concomitant use of ticagrelor and ritonavir)
* Patients on concomitant treatment with an anticoagulant agent (Vitamin-K antagonists or novel oral anticoagulants such as rivaroxaban, dabigatran or apixaban)
* Planned surgery within 12 coming months
* Patient under guardianship or curatorship
* Pregnancy or breastfeeding
* Inability to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2468 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Rate of combinated major and minor bleeding events (BARC 2 to 5 BARC) | From randomization (1-3months after inclusion) to 1year after inclusion
  the occurrence of major or minor bleeding events between randomization to one of the de-escalation strategies and 1 year after index ACS defined according to the Bleeding Academic Research Consortium (BARC) classification as type 2 to 5

SECONDARY OUTCOMES:
Rate of major adverse cardiovascular events | From randomization to de-escalation (1-3months) to 1year
  major adverse cardiovascular events defined as follow and in the following hierarchical order:
  * Death or myocardial infarction or stroke or stent thrombosis (key secondary)
  * Death or Myocardial infarction
Rate of major bleeding events | randomization to de-escalation (1-3months) to 1year
  the occurrence of major bleeding events between randomization to one of the de-escalation strategies and 1 year after index ACS defined according to the Bleeding Academic Research Consortium (BARC) classification
Rate of minor bleeding events | randomization to de-escalation (1-3months) to 1year
  the occurrence of minor bleeding events between randomization to one of the de-escalation strategies and 1 year after index ACS defined according to the Bleeding Academic Research Consortium (BARC) classification

CONTACTS AND LOCATIONS:
Overall Officials: Michel ZEITOUNI, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Pitié Salpetrière, Paris, IDF, France